CLINICAL TRIAL: NCT07336641
Title: LANDSCAPE - Demographic Characteristics and Treatment Profiles of Patients Affected by Inflammatory Skin Diseases (Psoriasis, Atopic Dermatitis, Alopecia Areata, Vitiligo, Hidradenitis Suppurativa) in Italian Clinical Practice
Brief Title: LANDSCAPE: Demographics and Treatment Patterns of Patients With Immune-Mediated Inflammatory Skin Diseases in Italian Clinical Practice
Acronym: LANDSCAPE
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione ISIDE (Other)
Responsible Party: Sponsor
Other Study IDs: ISIDE-LANDSCAPE-2025-001
Record Dates: First submitted 2025-12-30; First posted 2026-01-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis; Atopic Dermatitis; Vitiligo; Alopecia Areata; Hidradenitis Suppurativa
Keywords: Registry; Real-World Evidence; Treatment Patterns; Dermatology; Italy
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic; Vitiligo; Alopecia Areata; Hidradenitis Suppurativa | interventions — Biological Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Psoriasis Cohort: Adult patients (≥18 years) diagnosed with moderate-to-severe psoriasis according to clinical criteria, treated with systemic conventional and/or biologic therapies at participating Italian dermatology centers. No intervention is administered; data are collected retrospectively from medical records.
  Interventions: Drug: Conventional Systemic Therapies; Drug: Biologic Therapies
- Atopic Dermatitis Cohort: Adult patients (≥18 years) diagnosed with moderate-to-severe atopic dermatitis, treated with systemic conventional and/or biologic therapies at participating Italian dermatology centers. No intervention is administered; data are collected retrospectively from medical records.
  Interventions: Drug: Conventional Systemic Therapies; Drug: Biologic Therapies
- Alopecia Areata Cohort: Adult patients (≥18 years) diagnosed with alopecia areata, treated with systemic therapies at participating Italian dermatology centers. No intervention is administered; data are collected retrospectively from medical records.
  Interventions: Drug: Conventional Systemic Therapies; Drug: Biologic Therapies
- Vitiligo Cohort: Adult patients (≥18 years) diagnosed with vitiligo, treated at participating Italian dermatology centers. No intervention is administered; data are collected retrospectively from medical records.
  Interventions: Drug: Conventional Systemic Therapies; Drug: Biologic Therapies
- Hidradenitis Suppurativa Cohort: Adult patients (≥18 years) diagnosed with hidradenitis suppurativa, treated with systemic conventional and/or biologic therapies at participating Italian dermatology centers. No intervention is administered; data are collected retrospectively from medical records
  Interventions: Drug: Conventional Systemic Therapies; Drug: Biologic Therapies

INTERVENTIONS:
Drug: Conventional Systemic Therapies — Retrospective observation of conventional systemic treatments prescribed in routine clinical practice, including but not limited to methotrexate, cyclosporine, acitretin, and other conventional agents. No drugs are administered as part of this study; treatment data are collected from existing medical records.
Drug: Biologic Therapies — Retrospective observation of biologic treatments prescribed in routine clinical practice, including but not limited to TNF-α inhibitors, IL-17 inhibitors, IL-23 inhibitors, IL-4/IL-13 inhibitors, and JAK inhibitors. No drugs are administered as part of this study; treatment data are collected from existing medical records.

SUMMARY:
This multicenter retrospective observational registry study will collect existing clinical data from Italian centers to describe epidemiology, treatment patterns, clinical evolution, safety, and comorbidities in patients aged 12 years and older with psoriasis, atopic dermatitis, vitiligo, alopecia areata, or hidradenitis suppurativa.

DETAILED DESCRIPTION:
LANDSCAPE is a non-interventional, multicenter, retrospective disease registry based on routinely collected clinical data (electronic health records and available medical documentation) from participating Italian centers. Data will cover the period January 2016 to December 2025. The registry will support real-world evaluation of treatment patterns, effectiveness and safety outcomes, disease severity scores, persistence/switching, and associated comorbidities across psoriasis, atopic dermatitis, vitiligo, alopecia areata, and hidradenitis suppurativa. Data will be pseudonymized prior to entry into the EDC system. Patients who exercise the opt-out right will not be included.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of psoriasis, atopic dermatitis, vitiligo, alopecia areata, or hidradenitis suppurativa.
2. Age 12 years or older at the first recorded visit.
3. Eligible for or treated with systemic therapies.
4. At least one documented visit during January 2016 to December 2025.
5. No opt-out exercised.

Exclusion Criteria:

1. Opt-out exercised.
2. Medical records with insufficient data.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with inflammatory skin diseases (psoriasis, atopic dermatitis, alopecia areata, vitiligo, hidradenitis suppurativa) followed at approximately 25 dermatology centers across Italy. The study population reflects real-world clinical practice, including patients managed in both academic and community dermatology settings within the Italian National Health Service (Servizio Sanitario Nazionale). Data are extracted retrospectively from routine medical records.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Patient Distribution by Disease Type | January 2016 to December 2025
  Number and proportion of patients in each disease cohort (psoriasis, atopic dermatitis, alopecia areata, vitiligo, hidradenitis suppurativa).
Age at Treatment Initiation | January 2016 to December 2025
  Mean age (years) at first systemic treatment initiation, reported by disease cohort.
Sex Distribution | January 2016 to December 2025
  Proportion of male and female patients (percentage) by disease cohort.

SECONDARY OUTCOMES:
Treatment Patterns and Therapeutic Sequences | January 2016 to December 2025
  Description of systemic treatment utilization patterns, including conventional and biologic therapies, lines of therapy, treatment switches, and reasons for discontinuation.
Disease Severity Assessment Over Time | January 2016 to December 2025
  Evaluation of disease severity measures as recorded in routine clinical practice, including PASI for psoriasis, EASI/IGA for atopic dermatitis, SALT for alopecia areata, and Hurley staging for hidradenitis suppurativa.
Treatment Persistence and Drug Survival | January 2016 to December 2025
  Analysis of treatment duration and persistence rates for systemic therapies in real-world clinical practice

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Clinico Humanitas - Dermatology Unit, Rozzano, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be shared due to data protection requirements under GDPR (EU 2016/679) and Italian privacy legislation. Aggregate anonymized results will be published in peer-reviewed journals and presented at scientific conferences.